CLINICAL TRIAL: NCT07029087
Title: The Effect of Pudendal Block on Postoperative Analgesia in Urogynecological Surgeries
Brief Title: The Effect of Ultrasound Guided Pudendal Block on Postoperative Analgesia in Urogynecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Azime Bulut, Associate professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Azime Bulut
Record Dates: First submitted 2025-05-05; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Urinary Incontinence
Keywords: postoperative analgesia; pudendal block; urogynecological surgery
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Randomized-controlled, double-blind study
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal (Experimental): We performed pudendal nerve block by using ultrasound at the end of the surgery. All patients were operated under spinal anesthesia. After surgery we followed up the hemodynamic changes and VAS values at different time points.
  Interventions: Procedure: Pudendal Nerve Block
- Control (No Intervention): All patients were operated under spinal anesthesia. After surgery we followed up the hemodynamic values and VAS scores at different time points.

INTERVENTIONS:
Procedure: Pudendal Nerve Block — Pudendal nerve blocks are often preferred as an initial diagnostic and therapeutic method for chronic pelvic pain caused by pudendal neuralgia due to nerve entrapment. Additionally, the pudendal nerve block is a widely used regional anesthesia technique in gynecologic, obstetric, and anorectal procedures . It is particularly applied to provide perineal anesthesia during the second stage of vaginal delivery, vaginal repairs, and obstetric procedures including anorectal surgeries such as hemorrhoidectomy . Pudendal nerve blocks can effectively anesthetize the posterior perineum, anus, lower vagina, vulva/scrotum, and penis.
  Arms: Pudendal

SUMMARY:
Stress urinary incontinence (SUI) is one of the most common problems encountered in gynecology outpatient clinics and affects approximately 4% to 35% of women. Although it is a medical condition, it also negatively impacts women's quality of life, making successful treatment of this condition particularly important from the patient's perspective. Additionally, overactive bladder and pelvic organ prolapse are frequently seen, especially in older women, and surgical procedures such as transobturator tape (TOT), cystocele repair, and rectocele repair are commonly performed to address these issues. In general, any type of surgical procedure in elderly patients is considered to carry higher risks compared to the younger population. Specifically, in prolapse surgeries, longer hospital stays and higher rates of perioperative complications have been reported compared to younger patients . Moreover, postoperative pain is a significant barrier to the resumption of daily activities.

The innervation of the perineal portion of the pelvic floor muscles is provided by the pudendal nerve, which originates from the ventral roots of sacral segments S2 to S4. Pudendal nerve blocks are often preferred as an initial diagnostic and therapeutic method for chronic pelvic pain caused by pudendal neuralgia due to nerve entrapment. Additionally, the pudendal nerve block is a widely used regional anesthesia technique in gynecologic, obstetric, and anorectal procedures . It is particularly applied to provide perineal anesthesia during the second stage of vaginal delivery, vaginal repairs, and obstetric procedures including anorectal surgeries such as hemorrhoidectomy . Pudendal nerve blocks can effectively anesthetize the posterior perineum, anus, lower vagina, vulva/scrotum, and penis.

In this study, the investigators aimed to demonstrate the effectiveness of the pudendal nerve block in achieving postoperative analgesic control during urogynecological surgeries such as TOT, cystocele, and rectocele repairs, and thereby facilitating an earlier return to daily activities.

DETAILED DESCRIPTION:
The study was planned to be conducted prospectively, in a randomized and controlled manner on female patients who were scheduled for elective urogynecological surgery in the obstetrics operating room of Giresun Women's and Children's Hospital. Written and verbal informed consent will be obtained from all patients who agree to participate in the study. Group allocation will be determined using a randomization method via sealed opaque envelopes. The patients' age, height, weight, and American Society of Anesthesiologists (ASA) physical status classification will be recorded.

All patients will receive spinal anesthesia before surgery in the obstetrics operating room. At the end of the surgery, patients in the block group will undergo pudendal nerve block under ultrasound guidance. For the block procedure, aseptic preparation will be performed on the perineal area of the patient in the lithotomy position. A 21-gauge, 100 mm Stimuplex peripheral nerve block needle will be used. A linear ultrasound probe will be placed on the perineum at the 3 and 9 o'clock positions relative to the anus to visualize the ischial tuberosity. The needle will be inserted in an out-of-plane approach, medially to the ischial tuberosity, to reach the area between the sacrotuberous and sacrospinous ligaments. A total of 10 ml of 0.25% plain bupivacaine, diluted with isotonic solution, will be administered bilaterally.

Postoperative pain assessments using the Visual Analog Scale (VAS) will be performed at 2, 4, 6, 12, 24, and 48 hours in both the block and control groups. If a patient reports a VAS score greater than 4, intramuscular diclofenac sodium will be administered and recorded. Additionally, the time at which patients can sit without pain, the time to return to daily activity, and length of hospital stay will also be documented.

ELIGIBILITY:
Inclusion Criteria: >18 years ASA I-II scores Clinical diagnosis of urinary incontinence The patients with consent to be included in the study - Exclusion Criteria: Patients who suffer from chronic pain Patients using regular analgesic drugs Pregnant patients Allergic reactions to local anesthetics ASA III and over patients Need for general anesthesia

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators performed the pudendal nerve block to the patients who operated for urinary incontinence.
Enrollment: 58 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 24 hours after surgery
  The primary endpoint was the postoperative pain on the visual analogue scale (VAS) at 24 h. The investigators evaluated the pain intensity by using the VAS, where 0 indicated no pain and 10 represented the worst imaginable pain.

SECONDARY OUTCOMES:
Length of hospital stay | 14 days after surgery
  Length of hospital stay: The number of days that stayed in hospital
The time of sitting without pain | 24 hours after surgery
  The investigators recorded how many hours after the surgery the patients were able to sit without pain.
Analgesic need | 24 hours after surgery
  Analgesic consumption: Total amount of analgesic need during first 24 hours on postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Azime Bulut, Assoc.Prof., Principal Investigator — Giresun University
Locations (1):
- Giresun Training and Research Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators don't have any consent or permission for sharing the data.

REFERENCES:
- [Background] Naja Z, El-Rajab M, Al-Tannir M, Ziade F, Zbibo R, Oweidat M, Lonnqvist PA. Nerve stimulator guided pudendal nerve block versus general anesthesia for hemorrhoidectomy. Can J Anaesth. 2006 Jun;53(6):579-85. doi: 10.1007/BF03021848. PMID 16738292
- [Background] He J, Zhang L, Li DL, He WY, Xiong QM, Zheng XQ, Liao MJ, Wang HB. Ultrasound-Guided Pudendal Nerve Block Combined with Propofol Deep Sedation versus Spinal Anesthesia for Hemorrhoidectomy: A Prospective Randomized Study. Pain Res Manag. 2021 Feb 26;2021:6644262. doi: 10.1155/2021/6644262. eCollection 2021. PMID 33727997
- [Background] Di Giuseppe M, Saporito A, La Regina D, Tasciotti E, Ghielmini E, Vannelli A, Pini R, Mongelli F. Ultrasound-guided pudendal nerve block in patients undergoing open hemorrhoidectomy: a double-blind randomized controlled trial. Int J Colorectal Dis. 2020 Sep;35(9):1741-1747. doi: 10.1007/s00384-020-03630-x. Epub 2020 May 30. PMID 32474710